CLINICAL TRIAL: NCT05411107
Title: Phase II Trial of Oral Iloprost for the Precision Chemoprevention of Lung Cancer
Brief Title: Oral Iloprost for the Prevention of Lung Cancer In Former Smokers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Agent is not available
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2022-04698; NCI-2022-04698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI21-08-01 (Other: Northwestern University); NWU21-08-01 (Other: DCP); P30CA060553 (NIH); UG1CA242643 (NIH)
Record Dates: First submitted 2022-06-08; First posted 2022-06-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Bronchial Epithelial Dysplasia; Chronic Obstructive Pulmonary Disease; Lung Carcinoma; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Tobacco-Related Carcinoma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms | interventions — Specimen Handling; Bronchoscopy; Iloprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (iloprost) (Experimental): Patients receive Iloprost PO BID for a 180 days in the absence of unacceptable toxicity. Patients undergo bronchoscopy with biopsies and brushings at day 180.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bronchial Brush Biopsy; Procedure: Bronchoscopy; Drug: Iloprost; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for a 180 days in the absence of unacceptable toxicity. Patients undergo bronchoscopy with biopsies and brushings at day 180.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bronchial Brush Biopsy; Procedure: Bronchoscopy; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of sputum sample
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bronchial Brush Biopsy — Undergo bronchial brush biopsy
  Other Names: bronchial brushing
Procedure: Bronchoscopy — Undergo bronchoscopy
Drug: Iloprost — Given PO
  Other Names: Ciloprost; Iloprost Clathrate; Ventavis; ZK 36374
  Arms: Arm I (iloprost)
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests whether oral iloprost works in preventing lung cancer (chemoprevention) in former smokers. Oral iloprost has previously been shown to reduce abnormal lung cells in former smokers, suggesting a clinically significant impact on lung cancer risk. The use of oral iloprost may help keep cancer from forming and reduce abnormal cells in the lung in order to lower the risk of developing lung cancer in former smokers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I.To determine if oral iloprost, starting at 50 ug twice daily (BID) and increased monthly to a final dose of 150 ug BID as tolerated, compared to placebo for 6 months is effective in reducing endobronchial dysplasia in former smokers who have mild or worse dysplasia on an endobronchial biopsy at baseline bronchoscopy.

SECONDARY OBJECTIVES:

I. To determine if treatment with oral iloprost compared to placebo results in a change in average dysplasia (over all sites of mild or greater dysplasia).

II. To determine safety of treatment with oral iloprost.

EXPLORATORY OBJECTIVES:

I. To determine if treatment with oral iloprost compared to placebo results in a change in response rate defined as >= 1 point reduction in maximum dysplasia.

II. To determine if the in vitro differentiation response of bronchial epithelial cell progenitors cultured at the air liquid interface is predictive of the in vivo response of dysplasia improvement (to be done only in participants recruited in Colorado).

III. To determine if treatment with oral iloprost compared to placebo results in a decrease in the volume of pure ground glass opacities (GGOs) on chest computed tomography (CT).

IV. To determine if treatment with oral iloprost compared to placebo increases peripheral lung epithelial progenitor counts, measured by organoid formation in a three dimensional culture system seeded from distal airway brushings (to be done only in participants recruited in Colorado).

V. To determine if oral iloprost reduces the incidence of lung cancer compared to placebo.

VI. To evaluate the ability of 3-dimensional morphologic analysis of expectorated sputum by LuCED compared to standard sputum cytopathology to predict endobronchial dysplasia and measure response to iloprost.

VII. To evaluate histologic response by alternative criteria.

OUTLINE: Patients are randomized in 1 of 2 arms.

ARM I: Patients receive iloprost orally (PO) BID for a 180 days in the absence of unacceptable toxicity. Patients undergo bronchoscopy with biopsies and brushings at day 180.

ARM II: Patients receive iloprost placebo PO BID for a 180 days in the absence of unacceptable toxicity. Patients undergo bronchoscopy with biopsies and brushings at day 180.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be former smokers (> 12 months abstinent and confirmed by serum cotinine) with at least a 30 pack-year cigarette history who are at high risk for the development of lung cancer with at least one of the following:

  * Stage I or II lung cancer survivors, surgically treated with curative intent, who have remained disease free for > 12 months. Participants may have been treated with adjuvant chemotherapy or targeted therapy [(e.g. Osimertinib for epidermal growth factor receptor (EGFR) mutation)], if appropriate, provided they are > 12 months from the last systemic adjuvant therapy dose.
  * Patients with chronic obstructive pulmonary disease (COPD), defined as either airflow obstruction (forced expiratory volume in 1 second [FEV1]/forced vital capacity [FVC] < 0.70) on spirometry or emphysema (as commented on in a Radiology report) on CT scan.
  * Patients who display a ground glass opacity (GGO) on CT with a largest diameter =< 10 mm and >= 4 mm on axial imaging. The GGO must either be documented to have remained the same size or slowly progressing, but not regressing, over a 6-month period of observation by serial CT scan such that further workup beyond observation is not planned. A solid component of =< 1/3 of the axial diameter may be present, providing the treating physician(s) do not plan on workup for resection within the next 6 months, taking both the character of the lesion and its rate of growth into consideration.
  * Patients who have had a previous endobronchial biopsy with mild World Health Organization (WHO) score 4 or greater dysplasia
* Participants must be able to safely undergo bronchoscopy in the judgement of the investigator
* Participants must have a biopsy showing mild (grade 4 on WHO score) or greater dysplasia on the baseline bronchoscopy
* Participants must be at least 50 years old. Because no dosing or adverse event (AE) data are currently available on the use of iloprost in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (ULN)
* Creatinine =< 2.0 mg/dl
* The effects of iloprost on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because prostacyclins are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* The use of any tobacco product or inhalational nicotine delivery device in the past year
* Taking any anticoagulant agent with the exception of aspirin
* Taking any antiplatelet agent
* Receiving any other investigational agents or the previous use of iloprost
* Participants may not have received radiation therapy directed to the thorax or head and neck or immunotherapy, including checkpoint inhibitors
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to iloprost
* A requirement of supplemental oxygen (O2) of >= 4 liter/minute to maintain an oxygen saturation of >= 90% at rest
* A biopsy on baseline bronchoscopy with a dysplasia score of 7 or 8 (carcinoma in situ or invasive cancer)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because iloprost is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with iloprost breastfeeding should be discontinued if the mother is treated with iloprost.
* Due to the risk for hypotension due to vasodilator effect of iloprost, participants must not have a blood pressure < 95 mm Hg systolic
* Participants must not have a current or prior invasive cancer within the past 12 months. History of the following cancers, curatively treated by surgery or locally ablative means, at any time prior to screening is allowed: non-melanoma skin cancer and cervical carcinoma in situ. Participants with prostate cancer undergoing active surveillance are allowed.
* Participants being treated with hormonal or immune therapies, including intravesicular bacillus calmette-guerin (BCG), are excluded
* Survivors of curatively treated stage III non-small cell lung cancer (NSCLC) or any stage lung small cell carcinoma (SCLC) are excluded
* Patients with known metastatic cancer of any kind are excluded
* Participants with known underlying bleeding disorders are excluded

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in numerical grade of the worst (highest grade on the WHO scale) dysplastic lesion per subject on bronchoscopy | Baseline to 6 month follow up
  Histologic response is the mean change between baseline and 6 month follow up bronchoscopy in the numerical grade of the worst (highest grade on the World Health Organization [WHO] scale) dysplastic lesion per subject. Will be analyzed using a linear regression models with post-treatment worst grade dysplasia as the outcome variable, and treatment arm (iloprost and placebo) and baseline worst grade dysplasia as predictors.

SECONDARY OUTCOMES:
Change in the average WHO score of all biopsy sites with a baseline score of 4 or greater | Up to 6 months
  Will be assessed using bronchial biopsies according to the WHO grading system, where 1 is normal and 8 is invasive cancer.
Incidence of adverse events with oral iloprost | From first dose to end of study, assessed up to 6 months
  Safety will be assessed according to a comparison of adverse events (AEs) between iloprost and placebo participants. Descriptive statistics (frequency, percent) will be used to summarize participants' worst grade toxicity for each AE type. AE rates will be compared between treatment arms using Fisher's exact test since AE rates are expected to be low.

OTHER OUTCOMES:
Treatment response rate | Up to 6 months
  Treatment response will be defined as >= 1 point reduction in maximum dysplasia at end of treatment, and response rates will be compared between arms using a chisquared test.
In vitro response of bronchial epithelial progenitor cells cultured at the air-liquid interface | Up to 6 months
  Will compare the ability of iloprost exposure versus vehicle, to restore differentiation to ciliated and mucus secreting cells. This will then be compared to the in vivo response of the dysplastic lesion at the same biopsy site to iloprost or placebo as a potential predictive biomarker. This endpoint will only be assessed in biopsies from participants enrolled in Colorado.
Change in glass opacity (GGOs) volume | Up to 6 months
  Changes will be summarized using descriptive statistics, and a two-sample t-test or the Wilcoxon rank-sum test will be used to compare changes between the two arms.
Organoid formation | Up to 6 months
  Peripheral lung epithelial progenitor cells will be assessed for organoid formation in a three dimensional culture system before and after treatment with iloprost or placebo.The progenitor cells assay will be used to predict whether a participant will respond to iloprost (yes/no).
Morphologic analysis of expectorated sputum by LuCED | Up to 6 months
  Will evaluate the ability of 3-dimensional morphologic analysis of expectorated sputum by LuCED compared to standard sputum cytopathology to predict endobronchial dysplasia and measure response to iloprost.
Histologic response by alternative criteria | Up to 6 months
  Bronchoscopic biopsies of standard and visually abnormal sites will be graded on the WHO scale of dysplasia and assigned numerical scores from 1 (normal) to 8 (invasive cancer). Each lesion will be classified as complete response, partial response, stable disease or progressive disease based on Lam et al. and each response rate will be calculated on a per-site and per-participant basis.

CONTACTS AND LOCATIONS:
Overall Officials: York E Miller, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm